# Statistical Analysis Plan I5B-MC-JGDR

A Phase 1b Study of Olaratumab, Doxorubicin and Ifosfamide in the Treatment of Patients With Advanced or Metastatic Soft Tissue Sarcoma

NCT03283696

Approval Date: 28-Aug-2017

# 1. Statistical Analysis Plan I5B-MC-JGDR: A Phase 1b Study of Olaratumab, Doxorubicin and Ifosfamide in the Treatment of Patients with Advanced or Metastatic Soft Tissue Sarcoma

#### **Confidential Information**

The information contained in this document is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries.

Note to Regulatory Authorities: this document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries..

#### Olaratumab (LY3012207) Soft Tissue Sarcoma

Study JGDR is a Phase 1b, multicenter, nonrandomized, open-label study of intravenous olaratumab (15 mg/kg on Days 1 and 8 or 20-mg/kg loading dose on Days 1 and 8 in Cycle 1 followed by 15 mg/kg on Days 1 and 8 of subsequent cycles) combined with doxorubicin (25 mg/m² on Days 1, 2, 3), ifosfamide (2.5 g/m² on Days 1, 2, 3, 4) and mesna (≥60% of ifosfamide dose on Days 1, 2, 3, 4) in 21-day cycles in the treatment of patients with advanced or metastatic soft tissue sarcoma. Patients will receive combination treatment for a maximum of 6 cycles followed by olaratumab as monotherapy until there is evidence of disease progression, death, intolerable toxicity, or other withdrawal criteria are met.

Eli Lilly and Company Indianapolis, Indiana USA 46285 Protocol I5B-MC-JGDR Phase 1b

Statistical Analysis Plan electronically signed and approved by Lilly on date provided below.

Approval Date: 28-Aug-2017 GMT

# 2. Table of Contents

| Section | | Page |
|---|---|---|
| Olaratu | cal Analysis Plan I5B-MC-JGDR: A Phase 1b Study of mab, Doxorubicin and Ifosfamide in the Treatment of with Advanced or Metastatic Soft Tissue Sarcoma | 1 |
| 2. Table o | of Contents | 2 |
| 3. Revisio | on History | 6 |
| 4. Study ( | Objectives | 7 |
| 4.1. Prin | nary Objective | 7 |
| 4.2. Seco | ondary Objectives | 7 |
| 4.3. Exp | loratory Objectives | 7 |
| 5. A Prior | ri Statistical Methods | 8 |
| 5.1. Sam | nple Size Determination | 8 |
| 5.2. Gen | eral Considerations | 8 |
| 5.2.1. | Populations | 8 |
| 5.2.2. | Definitions and Conventions | 8 |
| 5.3. Han | dling of Dropouts or Missing Data | 8 |
| 5.4. Mul | tiplicity adjustment | 8 |
| 5.5. Pati | ent Disposition | 9 |
| 5.6. Pati | ent Characteristics | |
| 5.6.1. | Demographics | |
| 5.6.2. | Baseline Disease Characteristics | |
| 5.6.3. | Historical Illnesses | |
| 5.6.4. | Prior Therapies | |
| 5.6.5. | Poststudy Treatment Discontinuation Therapies | |
| | comitant Therapy | |
| | ety Analyses | |
| | Extent of Exposure | |
| 5.8.2. | Dose-Limiting Toxicity and DLT-Equivalent Toxicities | |
| 5.8.3. | Adverse Events | |
| 5.8.4. | Deaths, Other Serious Adverse Events | 12 |
| 5.8.5. | Medical History Related to Infusion Related Reactions or Hypersensitivity | 12 |
| 5.8.6. | Clinical Laboratory Evaluation. | |
| 5.8.7. | Vital Signs and Other Physical Findings | |
| 5.8.8. | Electrocardiograms, Echocardiogram / Multiple Gated | 12 |
| 2.0.0. | Acquisition Scan | 12 |

| 5. | 9. Ef | ficacy Analyses | 13 |
|----|--------|--------------------------------------------------|----|
| | 5.9.1. | Objective Response Rate and Disease Control Rate | 13 |
| | 5.9.2. | Progression-Free Survival | 13 |
| | 5.9.3. | Duration of Response | 14 |
| | 5.9.4. | Overall Survival | 14 |
| 5. | 10. Su | ıbgroup Analyses | 15 |
| 5. | 11. Ph | narmacokinetics and Immunogenicity | 15 |
| 5. | 12. Bi | omarker Analysis | 15 |
| 5. | 13. De | evelopment Safety Update Report | 15 |
| 5. | 14. Cl | inical Trial Registry | 15 |
| 6. | Refer | rences | 17 |
| 7. | Appe | ndices | 18 |

| I5B-MC-JGDR Statistical Analysis Plan Version <sup>•</sup> |
|------------------------------------------------------------|
|------------------------------------------------------------|

| P | aq | е | 4 |
|---|----|---|---|

#### **Table of Contents**

| Table | | Page |
|---|---|---|
| Table JGDR.5.1. | Rules for Determining Date of Progression or Censor for | |
| Progression-F | ree Survival | 14 |

# **Table of Contents**

| Appendix | | Page |
|-------------|---------------------------------------------|------|
| Appendix 1. | List of Preferred Terms for AESI. | 19 |
| Appendix 2. | List of Preferred Terms for Consolidated AE | 25 |

# 3. Revision History

Statistical Analysis Plan (SAP) Version 1 was approved prior to the first visit when a subject receives study drug or any other protocol intervention.

# 4. Study Objectives

# 4.1. Primary Objective

The primary objective is to characterize the safety profile of olaratumab when given in combination with doxorubicin, ifosfamide and mesna and to determine the dosing regimen appropriate for a future Phase 2 study.

# 4.2. Secondary Objectives

The secondary objectives are:

- to evaluate the pharmacokinetics (PK) of olaratumab when combined with doxorubicin, ifosfamide and mesna
- to evaluate the immunogenicity of olaratumab when combined with doxorubicin, ifosfamide and mesna
- to document any antitumor activity of olaratumab when combined with doxorubicin, ifosfamide and mesna

# 4.3. Exploratory Objectives

The primary objective is to explore biomarkers related to, but not limited to tumor microenvironment, immune cells/immune functioning, mechanism of action of study drugs, platelet-derived growth factor receptor (PDGF), cancer-related pathways and disease state, and their association with demographics, disease state and clinical outcomes.

#### 5. A Priori Statistical Methods

### 5.1. Sample Size Determination

The sample size determination is described in Protocol I5B-MC-JGDR (JGDR), Section 10.1.

#### 5.2. General Considerations

# 5.2.1. Populations

The following population will be defined for this study:

**Safety population**: All enrolled patients who receive any quantity of study treatment, regardless of their eligibility for the study, will be included in the safety analysis. Safety evaluation will be performed based on the actual initial therapy a patient has received. Efficacy analysis will be performed on the safety population unless otherwise specified.

**DLT-evaluable population**: The DLT-evaluable population will include all enrolled patients who complete Cycle 1 or discontinue due to a DLT prior to completing Cycle 1.

#### 5.2.2. Definitions and Conventions

The **baseline value** is the last non-missing value observed prior to the first dose of study treatment.

The **study day** will be calculated as: assessment date – first dose date + 1 day if the assessment is done on or after the first dose day. If the assessment is done prior to the first dose day, study day will be calculated as assessment date – first dose date.

Date of first dose is defined as study Day 1.

One month is defined as 365/12 days.

Unless otherwise noted, **summaries of continuous variables** will include mean, median, standard deviation, minimum, and maximum. When appropriate, lower and upper quartiles will also be presented.

Unless otherwise noted, summaries of **categorical variables** will include the frequency and percentage (relative to the population being analyzed) of each category.

# **5.3.** Handling of Dropouts or Missing Data

With the exception of dates, missing data will not be imputed. The method of imputation for any dates that are imputed is described in the relevant sections.

# 5.4. Multiplicity adjustment

Multiplicity will not be adjusted.

#### 5.5. Patient Disposition

The number and percentage of patients entered into the study, treated in the study, as well as reasons for discontinuation from study treatment and reasons for discontinuation from study, will be summarized overall as well as by treatment cohort. A listing of patient disposition will also be provided.

Significant protocol violations that potentially compromise the data integrity and patients' safety will be summarized for safety population. These violations will include deviations that can be identified programmatically and those that can only be identified by the clinical research associate during monitoring. Significant protocol violations are described in the Trial Issue Management Plan within the study Trial Master File.

#### 5.6. Patient Characteristics

# 5.6.1. Demographics

Patient demographics will be summarized for safety population. Patient demographics will include country, age, sex, race, ethnicity, height, weight, and body surface area (BSA).

#### 5.6.2. Baseline Disease Characteristics

Eastern Cooperative Oncology Group (ECOG) performance status (PS), initial pathological diagnosis, basis for initial diagnosis, disease stage, histopathological grade, TNM stage and time since initial diagnosis will be summarized for safety population using descriptive statistics and listed in a data listing.

#### 5.6.3. Historical Illnesses

Historical illnesses are clinically relevant events in the past that ended before the screening visit. Historical illnesses (using Preferred Terms [PT] from the most current version of the Medical Dictionary for Regulatory Activities [MedDRA<sup>TM</sup>]) will be summarized.

# 5.6.4. Prior Therapies

Prior radiotherapy, surgery, systemic and locoregiojnal therapy will be summarized. Prior radiotherapy will be categorized by reason (neoadjuvant, adjuvant, neoadjuvant plus adjuvant, advanced/metastatic) for the regimen and prior surgery will be categorized by intent (curative, palliative). Prior systemic and locoregiojnal therapy will be categorized by treatment intent (curative, palliative) and setting (neoadjuvant, adjuvant, locally advanced, metastatic). Frequency of each specific therapy will be tabulated within each type of regimen and reason for regimen.

# 5.6.5. Poststudy Treatment Discontinuation Therapies

Therapies received following study treatment discontinuation will be summarized overall and by type of therapy.

#### 5.7. Concomitant Therapy

Concomitant medications including indication for use (primary study condition, AE or medical history event, prophylaxis) will be summarized and listed.

# 5.8. Safety Analyses

All safety analyses will be performed on the safety population within each cohort. Safety analyses will also be performed combining patients treated within the dose confirmatory phase with patients treated at the same dose level within the dose finding phase.

# 5.8.1. Extent of Exposure

Drug exposure, dose intensity, drug adjustments (dose omissions, interruptions, reductions) and dose delays for olaratumab, doxorubicin, ifosfamide and mesna will be summarized for all treated patients.

Drug exposure will include the following summaries:

- Number of cycles received per patient
- Duration on therapy: (date of last cycle Day 1 date of first dose +21)  $\div$  7, [weeks]
- Cumulative dose: sum of dose administered at each infustion per patient per compound, [mg]
- Weekly dose intensity: the actual cumulative amount of drug taken divided by the duration of treatment in weeks
  - Olaratumab: cumulative dose / last available weight / duration of therapy, [mg/kg/week]
  - Doxorubicin: cumulative dose / BSA derived using last available weight / duration of therapy, [mg/m²/week]
  - o Ifosfamide: cumulative dose / BSA derived using last available weight / duration of therapy, [mg/m²/week]
  - Mesna: cumulative dose / BSA derived using last available weight / duration of therapy, [mg/m²/week]
- Relative dose intensity: the actual amount of drug taken divided by the amount of drug prescribed times 100%, [%]

The summary of dose adjustments and delays will include the reason for adjustment or delays.

# 5.8.2. Dose-Limiting Toxicity and DLT-Equivalent Toxicities

The definition and derivation of the dose limiting toxicities (DLT) and the DLT-equivalent toxicities (DET) is specified in Protocol JGDR, Section 7.2.2.

DLT will be summarized and listed for DLT-evaluable population. DET will also be listed and summarized for safety population.

#### 5.8.3. Adverse Events

Adverse event (AE) severity grades will be assigned by the investigator using Common Terminology Criteria for Adverse Events (CTCAE) Version 4. AE verbatim text will be mapped by the sponsor or designee to corresponding terminology within MedDRA.

**Pre-existing conditions** are defined as any AEs that begin prior to the first dose of study drug.

**Treatment-emergent adverse event** (TEAE) are defined as any AE that occurred or worsened between the day of first dose and up to 30-day follow-up visit (or up to any time if serious and related to study treatment).

Comparisons of pre-existing conditions to on-treatment events at the low level term (LLT) level will be used in the treatment-emergent computation.

The following AE will be considered as **AE of special interest** (AESI) for the combination of olaratumab and doxorubicin, ifosfamide and mesna: infusion-related reactions (IRR), cardiac arrhythmias, cardiac dysfunction, encephalopathy, renal toxicity. PT for AESI are listed in **Appendix 1**. Categories of AESI may be modified as the understanding of the safety of the investigational drug increases. The final list of categories will be reported in the clinical study report (CSR).

Consolidated AE will include Abdominal Pain, Anemia, Fatigue, Hyperbilirubinaemia, Hypertension, Hypoalbuminaemia, Hypokalaemia, Hypomagnesaemia, Hyponatraemia, Hypoproteinemia, Intestinal Obstruction, Leukocytosis, Leukopenia, Lymphopenia, Mucositis, Neuropathy, neutropenia, Musculoskeletal pain, Rash, and Thrombocytopenia. Each consolidated AE contains PTs identified as clinically identical or synonymous. PT for consolidated AEs are listed in Appendix 2.

The following summaries and listings will be produced:

- Overview of AE
- Summary of TEAE by PT (any grade and Grade  $\geq 3$ )
- Summary of DLT
- Summary of DET
- Summary of TEAE by system organ class (SOC) and PT (any grade and Grade ≥ 3)
- Summary of TEAE by SOC and PT and maximum grade (1-5)
- Summary of treatment-emergent serious AE (SAE) by SOC and PT (any grade and Grade  $\geq$  3)
- Summary of AEs as reason for study treatment discontinuation by SOC and PT
- Summary of and listing of TEAE leading to dose delays, omissions, interruptions, reductions, treatment discontinuation, hospitalizations, transfusions

- Summary of treatment-emergent AESI (any grade and Grade  $\geq 3$ )
- Summary of treatment-emergent consolidated AE (any grade and Grade  $\geq 3$ )
- Listings of DLT, DET, SAE, TEAE, AESI

The TEAE and SAE summaries will be produced for all TEAE/SAEs and repeated for TEAE/SAE related to study treatment, where relationship of the AE to the study treatment will be assessed by the investigator (yes or no).

#### 5.8.4. Deaths, Other Serious Adverse Events

A summary of all deaths, including reasons for deaths, will be provided. All deaths, deaths on therapy, deaths within 30 days of discontinuation of study therapy, deaths on therapy or within 30 days of discontinuation of study therapy, and deaths after 30 days of discontinuation of study therapy will be summarized by reason for death. For deaths due to AE, the preferred term will be provided. In addition to the tabular summary, a by-patient listing of all deaths on study not attributed to study disease by the investigator will be provided.

# 5.8.5. Medical History Related to Infusion Related Reactions or Hypersensitivity

Summaries will be provided for prespecified medical history related to IRR or hypersensitivity for a patient and patient's first degree relatives.

# 5.8.6. Clinical Laboratory Evaluation

All relevant laboratory values will be graded according to CTCAE Version 4. Treatmentemergent changes will be summarized by the maximum postbaseline grade, and a shift table of baseline grade by maximum postbaseline grade will be produced. A listing will be provided with a flag for values outside of the laboratory normal range.

# 5.8.7. Vital Signs and Other Physical Findings

Actual values and changes from baseline for vital signs including temperature, blood pressure, respiratory and heart rate will be summarized by scheduled time point using descriptive statistics and listed. A summary of ECOG performance status at each scheduled time point will be provided.

# 5.8.8. Electrocardiograms, Echocardiogram / Multiple Gated Acquisition Scan

Electrocardiograms (ECG) findings that are considered to be a medical history condition or an AE will be summarized and listed.

Left ventricular ejection fraction (LVEF) results will be summsrised by scheduled time point.

Changes in LVEF will also be summarized including percentage of patients with LVEF decrease of  $\geq$ 10% and below the lower limit of normal, or an absolute decrease of 20%, or an absolute LVEF decreases to or below 40%.

#### 5.9. Efficacy Analyses

All efficacy analyses will be performed on the safety population to investigate antitumor activity within each cohort. This study is not designed to perform hypothesis testing on efficacy.

Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 will be applied as the primary criteria for assessment of tumor response. Local tumor imaging (investigator assessment with site radiological reading) will be used.

All time-to-event variables will be estimated using Kaplan-Meier method (Kaplan and Meier 1958) and summary statistics including median along with 95% CI as well as even-free rates (and 95% CI) at different time points will presented.

# 5.9.1. Objective Response Rate and Disease Control Rate

Objective response rate (ORR) and disease control rate (DCR) are summary measures of best overall response (BOR) as defined by RECIST. BOR is derived from time point responses. All time point responses observed while on study treatment and during the short-term follow-up period (but before the initiation of postdiscontinuation therapy) will be included in the derivation. Best overall response of complete response (CR) and partial response (PR) should be confirmed by repeated assessment at least 4 weeks following the initial observation. Each patient's BOR will categorized as CR, PR, stable disease (SD), PD, or not evaluable (NE). If appropriate, the best overall tumor response may be derived using all available lesion measurement data to confirm the investigator assessments.

ORR will be estimated by dividing the total number of responders (CR+PR) by the number of treated patients. DCR is defined as the number of patients with SD, confirmed PR or confirmed CR (CR+PR+SD) divided by the number of treated patients. The estimates of ORR and DCR will be reported with exact 95% confidence interval (CI) for each arm.

Individual changes in the tumor burden over time will be presented graphically by waterfall and spier plots within a tumor type.

# 5.9.2. Progression-Free Survival

Progression-free survival (PFS) is defined as the time from the date of first dose until the date of radiographic documentation of progression (as defined by RECIST) based on investigator assessment or the date of death due to any cause, whichever is earlier. It is calculated as date of progression / censor – date of first treatment + 1.

Table JGDR.5.1 lists rules for determining date of progression or censor for PFS.

Table JGDR.5.1. Rules for Determining Date of Progression or Censor for Progression-Free Survival

| Rule | Situation | Date of Progression or Censor | Outcome |
|---|---|---|---|
| 1 | No baseline tumor assessment | Date of first dose | Censored |
| 2 | No postbaseline assessments and no death | Date of first dose | Censored |
| 3 | No documented progression and no death (with a postbaseline tumor assessment) | Date of last adequate tumor assessment | Censored |
| 4 | Patient lost to follow-up (or withdrew consent from study participation) before documented progression or death | Date of last adequate tumor assessment | Censored |
| 5 | Documented progression | Date of documented progression. If a tumor assessment was done on multiple days, use the earliest date for that visit. | Progressed |
| 6 | Death without documented progression | Date of death | Progressed |
| 7 | Documented progression or death after missing ≥2 consecutive postbaseline tumor assessments | Date of last adequate tumor assessment before missed assessments or date of first treatment, whichever is later. | Censored |

Note: Progression-free survival and associated outcome is determined by the earliest of the dates above, if more than 1 situation applies. If there are multiple dates associated with 1 radiological tumor assessment, the assessment date will be set to the first date when the overall response is PD and the last date otherwise. A radiological tumor assessment is considered adequate if its response is among CR, PR, SD, or PD. Symptomatic deteriorations (that is, symptomatic progressions, which are not radiologically confirmed) will not be considered as disease progressions.

# 5.9.3. Duration of Response

The duration of response (DoR) time is defined only for responders (patients with a confirmed CR or PR). It is measured from the date of first evidence of CR or PR to the date of objective progression or the date of death due to any cause, whichever is earlier. For clarity, the start date should be determined by the initial assessment of CR or PR, not the date of confirmation of CR or PR. It is calculated as date of progression or death – date of first response evaluation of CR or PR + 1.

Duration of response (DoR) will be censored according to the same rules as PFS, with the addition of the following rule: if a patient begins postdiscontinuation therapy, DoR will be censored on the day of the last response evaluation prior to the initiation of postdiscontinuation therapy.

#### 5.9.4. Overall Survival

Overall survival (OS) is defined as the time from the date of first dose until the date of death due to any cause. If the patient is alive at the cutoff date for the analysis (or was lost to follow-up without a confirmed date of death), OS will be censored on the last date the patient was known to be alive.

#### 5.10. Subgroup Analyses

Subgroup analyses may be performed as deemed appropriate. The following analyses will be considered, depending on the number of patients within each subgroup:

- Safety analyses based on different infusion type of doxorubicin (intravenous route of administration over 60 minutes versus a 24-hour continuous infusion).
- Safety analyses related to cardiac toxicity based on subgroup of patients received dexrazoxane.
- Safety analyses related to urotoxicity based on different mesna dose levels.

# 5.11. Pharmacokinetics and Immunogenicity

A separate analysis plan will be provided for PK and immunogenicity analyses.

#### 5.12. Biomarker Analysis

The detailed biomarker analysis will be included in a separate biomarker analysis plan.

# 5.13. Development Safety Update Report

The following reports are needed for the Development Safety Update Report (DSUR):

- Exposure information
- Listing of subjects who died during the DSUR period
- Discontinuations due to AEs during the DSUR Period

# 5.14. Clinical Trial Registry

Additional analyses will be performed for the purpose of fulfilling the Clinical Trial Registry (CTR) requirements. Analyses provided for the CTR requirements include the following:

- Summary of AEs, provided as a dataset which will be converted to an XML file. Both SAEs and "Other" AEs are summarized by treatment group and by MedDRA Preferred Term.
- An AE is considered "Serious" whether or not it is a TEAE.
- An AE is considered in the "Other" category if it is both a TEAE and is not serious.
- For each SAE and "Other" AE, for each term and treatment group, the following are provided:
  - o the number of participants at risk of an event (if certain subjects cannot be at risk for some reason, for example, gender-specific AEs, then the number will be adjusted to only include the patients at risk)
  - o the number of participants who experienced each event term
  - o the number of events experienced.

- For each SAE, for each term and treatment group, the following are also provided for the EudraCT results submission:
  - o The number of occurrences (events) causally related to treatment
  - The total number of deaths
  - o The number of deaths causally related to treatment
- Consistent with www.ClinicalTrials.gov requirements, a threshold for frequency of "Other" AEs can be implemented rather than presenting all "Other" AEs. For example, "Other" AEs that occur in fewer than 5% of patients in any treatment group may not be included if a 5% threshold is chosen. The frequency threshold must be less than or equal to the allowed maximum of 5%.
- A participant flow will be created that will describe:
  - Number of participants per treatment arm. Screen failures do not need to be included. Number of participants who did not complete the study per treatment arm. This analysis will be based on study discontinuation, not treatment discontinuation.
  - o Reasons participants did not complete the study.

# 6. References

Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. *J Am Stat Assoc.* 1958;53:457-481.

# 7. Appendices

# **Appendix 1. List of Preferred Terms for AESI**

#### **AESI**

Cardiac Dysfunction

#### **Preferred Term**

Acute left ventricular failure

Acute pulmonary oedema

Acute right ventricular failure

Cardiac asthma

Cardiac failure

Cardiac failure acute

Cardiac failure chronic

Cardiac failure congestive

Cardiac failure high output

Cardiogenic shock

Cardiopulmonary failure

Cardiorenal syndrome

Chronic left ventricular failure

Chronic right ventricular failure

Cor pulmonale

Cor pulmonale acute

Cor pulmonale chronic

Ejection fraction decreased

Hepatic congestion

Hepatojugular reflux

Left ventricular failure

Low cardiac output syndrome

Neonatal cardiac failure

Obstructive shock

Pulmonary oedema

Pulmonary oedema neonatal

Right ventricular failure

Ventricular failure

Artificial heart implant

Atrial natriuretic peptide abnormal

Atrial natriuretic peptide increased

Brain natriuretic peptide abnormal

Brain natriuretic peptide increased

Cardiac cirrhosis

Cardiac index decreased

Cardiac output decreased

Cardiac resynchronisation therapy

Cardiac ventriculogram abnormal

Cardiac ventriculogram left abnormal

Cardiac ventriculogram right abnormal

Cardiomegaly

AESI Preferred Term

Cardio-respiratory distress Cardiothoracic ratio increased

Central venous pressure increased

Diastolic dysfunction Dilatation ventricular

Dyspnoea paroxysmal nocturnal

Heart transplant

Hepatic vein dilatation
Jugular vein distension
Left ventricular dysfunction

Myocardial depression Nocturnal dyspnoea

N-terminal prohormone brain natriuretic

peptide abnormal

N-terminal prohormone brain natriuretic

peptide increased

Oedema

Oedema due to cardiac disease

Oedema neonatal Oedema peripheral

Orthopnoea

Peripheral oedema neonatal Pulmonary congestion

Right ventricular dysfunction

Scan myocardial perfusion abnormal

Stroke volume decreased Systolic dysfunction Venous pressure increased

Venous pressure jugular abnormal Venous pressure jugular increased Ventricular assist device insertion

Ventricular dysfunction Ventricular dyssynchrony Chronotropic incompetence

Electrocardiogram repolarisation abnormality Electrocardiogram RR interval prolonged Electrocardiogram U-wave abnormality

Sudden cardiac death

Bradycardia Cardiac arrest Cardiac death

Cardiac telemetry abnormal Cardio-respiratory arrest Electrocardiogram abnormal

Electrocardiogram ambulatory abnormal

Cardiac Arrhythmias

#### AESI

#### **Preferred Term**

Electrocardiogram change

Heart rate abnormal

Heart rate decreased

Heart rate increased

Loss of consciousness

**Palpitations** 

Rebound tachycardia

Sudden death

Syncope

Tachycardia

Tachycardia paroxysmal

Bradyarrhythmia

Ventricular asystole

Accessory cardiac pathway

Adams-Stokes syndrome

Agonal rhythm

Atrial conduction time prolongation

Atrioventricular block

Atrioventricular block complete

Atrioventricular block first degree

Atrioventricular block second degree

Atrioventricular conduction time shortened

Atrioventricular dissociation

Bifascicular block

Brugada syndrome

Bundle branch block

Bundle branch block bilateral

Bundle branch block left

Bundle branch block right

Conduction disorder

Defect conduction intraventricular

Electrocardiogram delta waves abnormal

Electrocardiogram PQ interval prolonged

Electrocardiogram PQ interval shortened

Electrocardiogram PR prolongation

Electrocardiogram PR shortened

Electrocardiogram QRS complex prolonged

Electrocardiogram QT prolonged

Electrocardiogram repolarisation abnormality

Lenegre's disease

Long QT syndrome

Sinoatrial block

Trifascicular block

Ventricular dyssynchrony

Wolff-Parkinson-White syndrome

#### AESI Preferred Term

Nodal arrhythmia

Nodal rhythm

Sick sinus syndrome

Sinus arrest

Sinus arrhythmia

Sinus bradycardia

Wandering pacemaker

Arrhythmia

Heart alternation

Heart rate irregular

Pacemaker generated arrhythmia

Pacemaker syndrome

Paroxysmal arrhythmia

Pulseless electrical activity

Reperfusion arrhythmia

Withdrawal arrhythmia

Arrhythmia supraventricular

Atrial fibrillation

Atrial flutter

Atrial parasystole

Atrial tachycardia

Junctional ectopic tachycardia

Sinus tachycardia

Supraventricular extrasystoles

Supraventricular tachyarrhythmia

Supraventricular tachycardia

ECG P wave inverted

Electrocardiogram P wave abnormal

Retrograde p-waves

Anomalous atrioventricular excitation

Cardiac flutter

Extrasystoles

Tachyarrhythmia

Accelerated idioventricular rhythm

Cardiac fibrillation

Parasystole

Rhythm idioventricular

Torsade de pointes

Ventricular arrhythmia

Ventricular extrasystoles

Ventricular fibrillation

Ventricular flutter

Ventricular parasystole

Ventricular pre-excitation

Ventricular tachyarrhythmia

| AESI | Preferred Term |
|------|----------------|

Ventricular tachycardia

Encephalopathy Blurred vision

Coma Confusion

Extrapyramidal symptoms

Hallucinations Psychotic behavior

Seizures Somnolence

Urinary incontinence Allergic oedema

Anaphylactic reaction Anaphylactic shock Anaphylactoid reaction Anaphylactoid shock

Angioedema

Ciculatory collapse Circumoral oedema Conjunctival oedema Corneal oedema

Cytokine release syndrome Dialysis membrane reaction

Distributive shock Drug hypersensitivity Epiglottic oedema

Eye oedema
Eye swelling
Eyelid oedema
Face oedema
Gingival oedema
Gingival swelling
Gleich's syndrome
Hypersensitivity

Idiopathic urticaria Infusion related reaction

Kounis syndrome

Laryngeal oedema

Laryngotracheal oedema

Limbal swelling

Lip oedema

Lip swelling

Oculorespiratory syndrome

Oedema mouth

Oropharyngeal swelling

Palatal oedema

Infusion-related Reactions

AESI Preferred Term

Periobital oedema Pharyngeal oedema Scleral oedema

Shock

Swelling face Swollen tongue Tongue oedema Tracheal oedema

Type 1 hypersensitivity

Urticaria

Urticaria cholinergic Urticaria chronic Urticaria popular Acute renal failure

Renal toxicity: Nephrotoxicity

Acute renal failure
Aminoaciduria

Chronic renal failure Cylindruria Decrease in glomerular filtration rate

Enzymuria

Fanconi syndrome

Glycosuria

Increased serum creatinine

Phosphaturia Proteinuria Renal dysfunction

Tubular acidosis Tubulointerstitial nephritis

Hemorrhagic cystitis

Hematuria RBC in urine

Renal toxicity: Urotoxicity

#### List of Preferred Terms for Consolidated AE Appendix 2.

**Consolidated AE Preferred Term** Abdominal pain Abdominal pain

Abdominal pain lower

Abdominal pain upper

Anaemia Anaemia

Haemoglobin decreased

Red blood cell count decrease

Fatigue Asthenia

Hypoalbuminaemia

Fatigue

Blood bilirubin increased Hyperbilirubinaemia

Hyperbilirubinaemia

Hypertension Hypertension

> Blood pressure increased Blood albumin decreased

Hypoalbuminaemia

Hypokalaemia Blood potassium decreased

Hypokalaemia

Blood magnesium decreased Hypomagnesaemia

> Hypomagnesaemia Magnesium deficiency

Hyponatraemia Blood sodium decreased

Hyponatraemia

Hypoproteinemia Hypoproteinemia

Protein total decreased

Intestinal obstruction Gastrointestinal obstruction

Intestinal obstruction

Small intestinal obstruction

Leukocytosis Leukocytosis

White blood cell count increased

Leukopenia Leukopenia

White blood cell count decreased

Lymphocyte count decreased Lymphopenia

Lymphopenia

Mucositis Aphthous stomatitis

> Mucosal inflammation Oropharyngeal pain

**Stomatitis** 

Musculoskeletal pain Arthralgia

Back Pain

Bone Pain Flank Pain

Groin Pain

**Consolidated AE Preferred Term** 

Muscle Spasms

Musculoskeletal Chest Pain

Musculoskeletal Pain

Myalgia Neck Pain

Pain In Extremity Hypoaesthesia

Neuropathy

Neuropathy peripheral

Paraesthesia

Peripheral sensory neuropathy

Neutropenia Neutropenia

Neutrophil count decreased

Rash **Dermatitis** 

> Dermatitis acneiform Dermatitis allergic Dermatitis bullous

Rash

Rash follicular Rash generalised Rash macular Rash papular Rash pruritic Rash pustular

Thrombocytopenia Platelet count decreased

Thrombocytopenia

Leo Document ID = bcc6fdde-8d46-4c69-a893-34d6098e01e9

Approver: PPD

Approval Date & Time: 28-Aug-2017 12:24:08 GMT Signature meaning: Approved